CLINICAL TRIAL: NCT03533751
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study Investigating the Efficacy, Safety, and Pharmacokinetic Profile of ANB020 Administered to Adult Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Efficacy, Safety, and Pharmacokinetic Profile of Etokimab (ANB020) in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: ATLAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB020-005; 2018-000331-27 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-05-23 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
Keywords: ANB020; etokimab; eczema; moderate to severe
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received matching placebo to etokimab, administered subcutaneously (SC) every 4 weeks (Q4W) for up to 16 weeks.
  Interventions: Drug: Placebo
- Etokimab 20 mg SC Q4W (Experimental): Participants received etokimab 20 milligrams (mg) administered SC Q4W for up to 16 weeks.
  Interventions: Biological: Etokimab
- Etokimab 300 mg load + 150 mg SC Q8W (Experimental): Participants received a 300 mg loading dose of etokimab on Day 1 then 150 mg etokimab administered SC every 8 weeks (Q8W) for up to 16 weeks. At Weeks 4 and 12 participants received placebo.
  Interventions: Biological: Etokimab; Drug: Placebo
- Etokimab 300 mg load + 150 mg SC Q4W (Experimental): Participants received a 300 mg loading dose of etokimab on Day 1 then 150 mg etokimab administered SC Q4W for up to 16 weeks.
  Interventions: Biological: Etokimab
- Etokimab 600 mg load + 300 mg SC Q4W (Experimental): Participants received a 600 mg loading dose of etokimab on Day 1 then 300 mg etokimab administered SC Q4W for up to 16 weeks.
  Interventions: Biological: Etokimab

INTERVENTIONS:
Biological: Etokimab — Humanized monoclonal antibody, administered by subcutaneous injection
  Other Names: ANB020
  Arms: Etokimab 20 mg SC Q4W; Etokimab 300 mg load + 150 mg SC Q4W; Etokimab 300 mg load + 150 mg SC Q8W; Etokimab 600 mg load + 300 mg SC Q4W
Drug: Placebo — Administered by subcutaneous injection
  Arms: Etokimab 300 mg load + 150 mg SC Q8W; Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety, and pharmacokinetic (PK) profiles of multiple doses of etokimab in adult participants with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants must be 18 to 75 years of age, at the time of signing the informed consent.
2. Body mass index (BMI) of 18 to ≤ 35 kilogram per square meter (kg/m^2) at screening.
3. Clinically confirmed diagnosis of AD.
4. Eczema Area and Severity Index (EASI) score ≥ 16, body surface area (BSA) involvement ≥ 10%, and an Investigator's Global Assessment (IGA) score (5-point scale) ≥ 3 at baseline.
5. Participants with a history of inadequate response to topical treatment, use of systemic treatments to treat AD, and/or for whom topical treatments are otherwise medically inadvisable.
6. Daily use of non-medicated emollient for at least 7 days prior to baseline.

Exclusion Criteria:

1. Treatment with topical corticosteroids, topical calcineurin inhibitors, or crisaborole within 2 weeks before dosing.
2. Prior exposure to an anti-interleukin (IL)-33 antibody.
3. Exposure to an investigational or licensed or other anti T-helper 2 (Th2) type cytokine or cytokine receptor antagonist within 16 weeks or 5 half-lives, whichever is longer.
4. History of prior exposure to any investigational or biologic systemic treatment within 5 half lives of the screening or is currently enrolled in another clinical study.
5. Have received systemic treatment for AD (including systemic corticosteroids, immunosuppressants or immunomodulating drugs, or phototherapy or use of a tanning booth) within 4 weeks before screening.
6. History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Randazzo, MD, Study Director — AnaptysBio, Inc.
Locations (81):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Encino Research Group, Encino, California
  - Irvine Center for Clinical Research, Inc., Irvine, California
  - Clinical Science Institute, Santa Monica, California
  - Medical Research Center of Miami, Miami, Florida
  - Compass Research Main, Orlando, Florida
  - Moore Clinical Research Inc. - Brandon, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc., Albany, Georgia
  - Dermatologic Surgery Specialists, Macon, Georgia
  - Marietta Dermatology & The Skin Cancer Center - Marietta, Marietta, Georgia
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Midwest Allergy, Sinus and Asthma, SC, Normal, Illinois
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - DermResearch, PLLC, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Grekin Skin Institute - Warren, Warren, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - JDR Dermatology Research, Las Vegas, Nevada
  - The Dermatology Group, Verona, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Forest Hills Dermatology Group, Forest Hills, New York
  - SRG, New York, New York
  - DermResearch Center of New York, Stony Brook, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Coppell Allergy and Asthma PA, Coppell, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Center for Medical Research, Houston, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
- Canada (7):
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - ICLS Dermatology and Plastic Surgery, Oakville, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Le centre de Recherche en Dermatologie du Drummondville, Drummondville, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
- Czechia (6):
  - CCR Brno, s.r.o., Brno
  - CCR Czech, a.s., Pardubice
  - CLINTRIAL s.r.o., Prague
  - Dermatovenereology, Prague
  - Fakultni nemocnice v Motole, Prague
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem o.z., Ústí nad Labem
- Germany (13):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Ludwigs-Maximilians-Universitaet Muenchen, Munich, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Lower Saxony
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera gGmbH, Gera, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Praxis fuer Haut- und Geschlechtskrankheiten, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Poland (13):
  - ClinicMed Daniluk, Nowak Spółka Jawna, Bialystok
  - Centrum Badan Klinicznych P.I. House Sp. z o.o., Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne All-Med, Krakow
  - Dermoklinika, Lodz
  - NZOZ ALL-MED Centrum Medyczne Specjalistyczne Gabinety Lekarskie, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej "Med-Laser", Lublin
  - Centrum Medyczne Medyk, Rzeszów
  - Laser Clinic S.C., Szczecin
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Clinical Research Group Sp. z o.o., Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- United Kingdom (5):
  - MAC UK Neurosciences Ltd / MAC Clinical Research, Manchester, Greater Manchester
  - MAC UK Neuroscience Ltd / MAC Clinical Research Ltd, Cannock, Staffordshire
  - Ninewells Hospital, Dundee
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.anaptysbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 75 centers in the United States, United Kingdom, Canada, Czech Republic, Germany, and Poland. The study enrolled adults with moderate to severe atopic dermatitis (AD).
  The study included a treatment period of 16 weeks (Week 0 to 16) followed by a safety follow-up for 8 weeks (Week 16 to Week 24).
Pre-assignment Details: Participants were equally randomized on Day 1 to one of five treatment groups.
Groups:
- Etokimab 300 mg / 150 mg SC Q8W: Participants received a 300 mg loading dose of etokimab on Day 1 then 150 mg etokimab administered SC every 8 weeks (Q8W) for up to 16 weeks. At Weeks 4 and 12 participants received placebo.
- Etokimab 300 mg / 150 mg SC Q4W: Participants received a 300 mg loading dose of etokimab on Day 1 then 150 mg etokimab administered SC Q4W for up to 16 weeks.
- Etokimab 600 mg / 300 mg SC Q4W: Participants received a 600 mg loading dose of etokimab on Day 1 then 300 mg etokimab administered SC Q4W for up to 16 weeks.
Period: Overall Study
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Started | 60 | 61 | 61 | 60 | 60
Treated | 60 | 61 | 59 | 60 | 60
Completed | 41 | 36 | 39 | 40 | 37
Not Completed | 19 | 25 | 22 | 20 | 23
Not completed — Withdrawal by Subject | 12 | 6 | 11 | 9 | 10
Not completed — Adverse Event | 4 | 7 | 2 | 4 | 5
Not completed — Physician Decision | 0 | 2 | 1 | 2 | 1
Not completed — Sponsor Decision | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 7 | 6 | 4 | 3
Not completed — Use of any excluded/prohibited medications | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 2 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least 1 dose of etokimab or placebo.
Groups:
- Placebo: Participants received matching placebo to etokimab, administered SC Q4W for up to 16 weeks.
- Etokimab 20 mg SC Q4W: Participants received etokimab 20 mg administered SC Q4W for up to 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W | Total
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (15.92) | 40.1 (16.76) | 39.7 (14.38) | 38.9 (14.61) | 37.1 (14.78) | 39.0 (15.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 36 | 24 | 32 | 146
  Male | 31 | 36 | 23 | 36 | 28 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 8 | 8 | 7 | 44
  Not Hispanic or Latino | 50 | 49 | 51 | 50 | 53 | 253
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 2 | 3
  Asian | 5 | 2 | 0 | 0 | 6 | 13
  Black or African American | 6 | 9 | 10 | 4 | 6 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 49 | 48 | 46 | 55 | 45 | 243
  Other | 0 | 1 | 3 | 1 | 1 | 6
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] — EASI measures the extent and severity of atopic eczema based on assessments of 4 body regions: head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected and the severity (scored as none [0], mild [1], moderate [2], or severe [3]) for symptoms such as redness (erythema), thickness (induration, papulation, and edema), scratching (excoriation), and lichenification (lined skin) are assessed. Total score is calculated by summing the EASI scores of 6 symptoms across 4 body regions. The EASI score ranges from 0 (no disease) to 72 (worse disease). Population: The Full Analysis Set included all randomized participants who received at least 1 dose of etokimab or placebo and had Baseline and post-baseline EASI scores. Number of participants with evaluable data were included.
  units on a scale
    number analyzed (Participants) | 59 | 61 | 59 | 60 | 60 | 299
    (all) | 26.6 (11.45) | 29.8 (12.08) | 27.1 (10.38) | 32.2 (13.06) | 29.5 (12.19) | 29.1 (11.92)
Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) [Count of Participants; unit: Participants] — The vIGA-AD is a 5-point scale to evaluate AD severity:
  * 0: Clear - No inflammatory signs of AD (erythema, induration/papulation, lichenification, oozing/crusting);
  * 1: Almost clear - Barely perceptible erythema, induration/papulation, minimal lichenification;
  * 2: Mild - Slight but definite erythema, induration/papulation, or lichenification. No oozing/crusting;
  * 3: Moderate - Clearly perceptible erythema, induration/papulation, or lichenification. Oozing or crusting may be present;
  * 4: Severe - Marked erythema, induration/papulation, or lichenification. Oozing or crusting may be present.
  Participants
    Grade 0 (Clear) | 0 | 0 | 0 | 0 | 0 | 0
    Grade 1 (Almost clear) | 0 | 0 | 0 | 0 | 0 | 0
    Grade 2 (Mild) | 0 | 0 | 0 | 0 | 0 | 0
    Grade 3 (Moderate) | 49 | 36 | 43 | 43 | 38 | 209
    Grade 4 (Severe) | 10 | 25 | 16 | 17 | 22 | 90
    Missing | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 16 in Eczema Area and Severity Index (EASI) Score
Description: EASI measures the extent and severity of atopic eczema based on assessments of 4 body regions: head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected and the severity (scored as none [0], mild [1], moderate [2], or severe [3]) for symptoms such as redness (erythema), thickness (induration, papulation, and edema), scratching (excoriation), and lichenification (lined skin) are assessed. Total score is calculated by summing the EASI scores of 6 symptoms across 4 body regions. The EASI score ranges from 0 (no disease) to 72 (worse disease).
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Missing data were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
percent change | -49.38 (7.124) | -41.63 (6.707) | -55.70 (6.206) | -47.40 (6.091) | -44.56 (7.811)
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.4498, ANCOVA; The p-value was obtained using a mixed effect analysis of covariance (ANCOVA) model with treatment as fixed effect and Baseline EASI as covariate; Least Squares (LS) Mean Difference = 7.75, 95% CI 2-sided [-12.4066 to 27.8983], Standard Error of Mean 10.235 — Difference = Etokimab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.5010, ANCOVA; The p-value was obtained using a mixed effect ANCOVA model with treatment as fixed effect and Baseline EASI as covariate; LS Mean Difference = -6.32, 95% CI 2-sided [-24.7740 to 12.1262], Standard Error of Mean 9.390 — Difference = Etokimab - Placebo
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.8349, ANCOVA; [statistical method as in outcome 1, analysis 2]; LS Mean Difference = 1.97, 95% CI 2-sided [-16.6037 to 20.5476], Standard Error of Mean 9.454 — Difference = Etokimab - Placebo
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.6662, ANCOVA; [statistical method as in outcome 1, analysis 2]; LS Mean Difference = 4.82, 95% CI 2-sided [-17.1892 to 26.8275], Standard Error of Mean 11.154 — Difference = Etokimab - Placebo

2. Secondary Outcome: Number of Participants With a 50% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 50 Response) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 21 | 19 | 27 | 21 | 18
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.7992, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.4200 to 1.9509]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.2197, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.7570 to 3.3572]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.7197, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.5345 to 2.4774]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.6772, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.3910 to 1.8404]

3. Secondary Outcome: Number of Participants With a 75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 75 Response) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 10 | 10 | 14 | 12 | 11
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.9537, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.3922 to 2.6994]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.3316, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.6323 to 3.8895]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.5166, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.5331 to 3.4944]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.7426, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.4545 to 3.0223]

4. Secondary Outcome: Number of Participants With a 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90 Response) at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 3 | 5 | 7 | 7 | 2
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.4543, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.3998 to 7.7615]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.1874, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.6314 to 10.4827]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.1721, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 2.69, 95% CI 2-sided [0.6506 to 11.0814]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.6755, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline EASI as a covariate; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.1086 to 4.2141]

5. Secondary Outcome: Number of Participants Who Achieved a Reduction of ≥ 2 Points From Baseline in the Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) at Week 16
Description: The vIGA-AD is a static 5-point scale to evaluate AD severity globally:
  0: Clear - No inflammatory signs of AD (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Postinflammatory hyperpigmentation and/or hypopigmentation may be present
  1. Almost clear - Barely perceptible erythema, barely perceptible induration/papulation, and/or minimal lichenification. No oozing or crusting
  2. Mild - Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification. No oozing or crusting
  3. Moderate - Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification. Oozing and crusting may be present
  4. Severe - Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification. Disease is widespread in extent. Oozing or crusting may be present.
  Number of participants with ≥2 points reduction in vIGA-AD is presented.
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 8 | 7 | 8 | 10 | 9
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.6058, Regression, Logistic; Logistic regression model with treatment as fixed effect and baseline vIGA-AD score as covariate; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.2481 to 2.2543]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.9521, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline vIGA-AD score as a covariate; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.3356 to 2.7923]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.6905, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline vIGA-AD score as a covariate; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.4457 to 3.3878]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.9399, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline vIGA-AD score as a covariate; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.3671 to 2.9518]

6. Secondary Outcome: Number of Participants Who Achieved a vIGA-AD Response of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: vIGA-AD is static 5-point scale to evaluate AD severity globally: 0: Clear - No inflammatory signs of AD (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Postinflammatory hyperpigmentation and/or hypopigmentation may be present
  1. Almost clear - Barely perceptible erythema, barely perceptible induration/papulation, and/or minimal lichenification. No oozing or crusting
  2. Mild - Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification. No oozing or crusting
  3. Moderate - Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification. Oozing and crusting may be present
  4. Severe - Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification. Disease is widespread. Oozing or crusting may be present Participants who achieved vIGA-AD response of 0 (clear) or 1 (almost clear) are reported.
Time Frame: Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 5 | 5 | 6 | 8 | 6
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.7659, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline vIGA-AD score as covariate; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.3290 to 4.5268]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.6273, Regression, Logistic; Logistic regression model with treatment as fixed effect and baseline vIGA-AD score as covariate; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.3895 to 4.7760]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.2967, Regression, Logistic; Logistic regression model with treatment as fixed effect and baseline vIGA-AD score as covariate; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.5734 to 6.1879]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.5544, Regression, Logistic; Logistic regression model with treatment as fixed effect and baseline vIGA-AD score as covariate; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.4152 to 5.1476]

7. Secondary Outcome: Number of Participants Who Achieved a Reduction of ≥ 4 Points From Baseline in Weekly Averaged Peak Numerical Rating Scale (NRS) for Pruritus Score at Week 16
Description: Participants were asked to rate itch (pruritis) intensity at its worst (peak) during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch) in a daily electronic diary. Weekly average was calculated as the average of the 7 days before each visit.
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Participants with missing data were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants | 5 | 6 | 8 | 9 | 9
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.8600, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline peak weekly averaged NRS as covariate; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.3175 to 3.9513]
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.3222, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline peak weekly averaged NRS as covariate; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.5511 to 6.1214]
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.2564, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline peak weekly averaged NRS as covariate; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.6089 to 6.4310]
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.2912, Regression, Logistic; Logistic regression model with treatment as fixed effect and Baseline peak weekly averaged NRS as covariate; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.5806 to 6.1275]

8. Secondary Outcome: Percent Change From Baseline in Peak Weekly Averaged Numerical Rating Scale (NRS) for Pruritus Score at Week 16
Description: as for outcome 7
Time Frame: Baseline and Week 16
Population: Full Analysis Set with available data were analyzed. Missing data were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 56 | 58 | 52 | 54 | 54
percent change | -21.13 (5.964) | -22.30 (6.211) | -17.69 (6.530) | -30.39 (6.176) | -27.18 (6.192)
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.8927, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline weekly averaged peak NRS as covariate; LS Mean Difference = -1.17, 95% CI 2-sided [-18.2117 to 15.8686], Standard Error of Mean 8.679 — Difference = Etokimab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.7035, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline weekly averaged peak NRS as covariate; LS Mean Difference = 3.43, 95% CI 2-sided [-14.2767 to 21.1463], Standard Error of Mean 9.019 — Difference = Etokimab - Placebo
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.2819, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline weekly averaged peak NRS as covariate; LS Mean Difference = -9.27, 95% CI 2-sided [-26.1590 to 7.6237], Standard Error of Mean 8.608 — Difference = Etokimab - Placebo
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.4793, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline weekly averaged peak NRS as covariate; LS Mean Difference = -6.06, 95% CI 2-sided [-22.8452 to 10.7333], Standard Error of Mean 8.557 — Difference = Etokimab - Placebo

9. Secondary Outcome: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as extent of disease (0 [no disease]-102 [worst disease]). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 (none) to 18 (severe intensity). Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (itch: 0 [no itch] to 10 [worst imaginable itch] and sleeplessness: 0 [no sleeplessness] to 10 [worst imaginable sleeplessness]) (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 (no AD present) to 103.4 (worst).
Time Frame: Baseline and Week 16
Population: Full Analysis Set. Missing data were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
percent change | -37.99 (4.764) | -31.42 (4.605) | -39.22 (4.294) | -35.48 (4.401) | -31.23 (4.927)
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.3262, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline SCORAD as covariate; LS Mean Difference = 6.57, 95% CI 2-sided [-6.5723 to 19.7054], Standard Error of Mean 6.677 — Difference = Etokimab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.8465, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline SCORAD as covariate; LS Mean Difference = -1.23, 95% CI 2-sided [-13.7439 to 11.2782], Standard Error of Mean 6.366 — Difference = Etokimab - Placebo
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.6947, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline SCORAD as covariate; LS Mean Difference = 2.51, 95% CI 2-sided [-10.0587 to 15.0820], Standard Error of Mean 6.396
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.3288, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline SCORAD as covariate; LS Mean Difference = 6.76, 95% CI 2-sided [-6.8451 to 20.3626], Standard Error of Mean 6.909 — Difference = Etokimab - Placebo

10. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much). Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Full Analysis Set with available data were analyzed. Missing data were imputed using multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 59 | 60
units on a scale | -5.61 (0.946) | -5.35 (0.966) | -6.52 (0.945) | -6.05 (0.945) | -5.18 (1.036)
Statistical Analysis 1: Comparison: Placebo vs Etokimab 20 mg SC Q4W; Test type: Superiority; p = 0.8497, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline DLQI score as covariate; LS Mean Difference = 0.26, 95% CI 2-sided [-2.4081 to 2.9218], Standard Error of Mean 1.355 — Difference = Etokimab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q8W; Test type: Superiority; p = 0.5016, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline DLQI score as covariate; LS Mean Difference = -0.91, 95% CI 2-sided [-3.5636 to 1.7473], Standard Error of Mean 1.350 — Difference = Etokimab - Placebo
Statistical Analysis 3: Comparison: Placebo vs Etokimab 300 mg / 150 mg SC Q4W; Test type: Superiority; p = 0.7511, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline DLQI score as covariate; LS Mean Difference = -0.44, 95% CI 2-sided [-3.1670 to 2.2870], Standard Error of Mean 1.386 — Difference = Etokimab - Placebo
Statistical Analysis 4: Comparison: Placebo vs Etokimab 600 mg / 300 mg SC Q4W; Test type: Superiority; p = 0.7558, ANCOVA; Mixed effect ANCOVA model with treatment as fixed effect and Baseline DLQI score as covariate; LS Mean Difference = 0.43, 95% CI 2-sided [-2.3133 to 3.1824], Standard Error of Mean 1.396 — Difference = Etokimab - Placebo

11. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A treatment-emergent adverse event (TEAE) is any AE that started or worsened in severity on or after the date and time of the study drug administration. A serious adverse event (SAE) is as any untoward medical occurrence that, at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent disability/incapacity;
  * Was a congenital anomaly/birth defect.
Time Frame: From first dose to Week 24
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
Number analyzed (Participants) | 60 | 61 | 59 | 60 | 60
Participants
  Any TEAE | 38 | 40 | 41 | 42 | 43
  Serious TEAE | 1 | 2 | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: From first dose to Week 24
Description: Safety Analysis Set
Arm/Group | Placebo | Etokimab 20 mg SC Q4W | Etokimab 300 mg / 150 mg SC Q8W | Etokimab 300 mg / 150 mg SC Q4W | Etokimab 600 mg / 300 mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61 | 0/59 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/61 | 3/59 | 3/60 | 3/60
Other Adverse Events (participants affected / at risk) | 24/60 | 22/61 | 23/59 | 18/60 | 26/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Etokimab 20 mg SC Q4W (N=61) | Etokimab 300 mg / 150 mg SC Q8W (N=59) | Etokimab 300 mg / 150 mg SC Q4W (N=60) | Etokimab 600 mg / 300 mg SC Q4W (N=60)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Joint Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Exfoliative Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Eczema Herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Etokimab 20 mg SC Q4W (N=61) | Etokimab 300 mg / 150 mg SC Q8W (N=59) | Etokimab 300 mg / 150 mg SC Q4W (N=60) | Etokimab 600 mg / 300 mg SC Q4W (N=60)
Nasopharyngitis (Infections and infestations) | 4 | 4 | 5 | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 1 | 2 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 12 | 6 | 8 | 9
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3 | 5
Oral Herpes (Infections and infestations) | 0 | 0 | 3 | 2 | 1
Impetigo (Infections and infestations) | 1 | 0 | 3 | 0 | 0
Conjunctivitis (Infections and infestations) | 3 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 3 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03533751/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03533751/SAP_001.pdf